CLINICAL TRIAL: NCT01155531
Title: A Phase I, Single Center, Open Label, Intra Subject, Dose Escalation Study to Evaluate Safety and Tolerability of Sertraline Plus Telenzepine in Overweight Healthy Subjects
Brief Title: Safety & Tolerability of a Combination of Antidepressant and Peptic Ulcer Drug in Overweight Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THR-4450-C-401
Record Dates: First submitted 2010-06-22; First posted 2010-07-01 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Sertraline; Telenzepine; Decrease appetite; Reduce appetite; Lose weight
MeSH Terms: conditions — Obesity; Overweight; Anorexia; Weight Loss | interventions — Sertraline; telenzepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telenzepine - Group A (Experimental): Group A: No Sertraline; 0, 1, 2, 3 mg/day Telenzepine
  Interventions: Drug: Sertraline plus Telenzepine
- Sertraline plus Telenzepine - Group B (Experimental): Sertraline 50 mg/day; 0, 1, 2, 3 mg/day Telenzepine
  Interventions: Drug: Sertraline plus Telenzepine
- Sertraline plus Telenzepine - Group C (Experimental): Sertraline 50, 100 mg/day; 0, 1, 2, 3 mg/day Telenzepine
  Interventions: Drug: Sertraline plus Telenzepine
- Sertraline plus Telenzepine - Group D (Experimental): Sertraline 50, 100, 150 mg/day; 0, 1, 2, 3 mg/day Telenzepine
  Interventions: Drug: Sertraline plus Telenzepine

INTERVENTIONS:
Drug: Sertraline plus Telenzepine — oral sertraline tablets at 0, 50, 100, or 150/day plus oral telenzepine capsules at 0, 1, 2, or 3 mg/day for 7 days in each combination

SUMMARY:
The hypothesis of this study is that up to 150 mg of sertraline and up to 3 mg of telenzepine will be safe, tolerable, and have the effect of suppressing appetite, when taken in combination daily by mouth by healthy, overweight, adult men and women.

In this study, up to 12 people will be assigned to one of 4 groups: A, B, C, and D, and will receive 0, 50, 100, or 150 mg of sertraline per day. People in Groups B, C, or D will receive an initial dose of 50 mg sertraline. People in Groups C and D will receive an additional 50 mg of sertraline per week.

Up to 10 people from each group who were able to tolerate their sertraline dose for at least 5 days will begin taking 50 mg of sertraline plus doses of telenzepine that will increase from 1 mg to 2 mg to 3 mg over a 7-day period (they will receive each combination). On the day before they begin taking this combination of drugs, their appetite will be evaluated (on a visual scale of 0 to 100) before and after 3 meals.

The appetites of each person, assessed by the visual scale, will be evaluated on the last day of the period (Day 7) before and after 3 meals of each combination treatment, while they are staying in the research unit. The amount of food they eat will be determined.

Based on safety and tolerability assessments of individuals, and of the previous groups who received lower doses of the combination of drug, a decision will be made whether to further increase the dose of these drugs.

Since the appetites of each person will be evaluated on the last day of the period (Day 7) before and after 3 meals of each combination treatment, people in this study will stay in the research unit for approximately 2½ days, starting on Day 6 of their previous treatment, so appetite evaluations can be made on Day 7 after a fixed meal in the evening of Day 6. These people will continue the stay in the research unit when they begin each telenzepine dose increase, so a 24 hour safety observation may be made immediately after the increase.

After the final doses of telenzepine have been received, people in Groups C and D will continue to receive sertraline 50 mg per day for an additional 7 days or until the study physician decides when sertraline should be discontinued. People will return to the study unit for final visit, 2 weeks after they have received their last sertraline dose.

ELIGIBILITY:
Inclusion Criteria:

* In good health based on medical history, physical examination, ECG, routine laboratory tests, and BMI >/= 30 kg/m2 and </=30 40 kg/m^2.
* Males and females agree to use described birth control methods.
* Non-smoker.
* Willing and able to be confined to the clinical research facility.
* Willing and able to comply with the protocol and able to communicate with investigators.
* Able to comprehend and willing to provide written informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, or allergic disease (including drug allergies; patients with untreated, asymptomatic, seasonal allergies may be enrolled), surgical conditions, cancer or any other condition that might in the opinion of the investigator impair the ability of the subject to complete the study or significantly interfere with the absorption, distribution, metabolism, or excretion of the study drugs.
* Evidence or history of clinically significant psychiatric disease including major depression, mania, or hypomania, and history of suicide attempts or suicidal ideation. Subjects with a Beck Depression Inventory-II (BDI-II) score >13 at screening are excluded.
* Clinically relevant abnormal findings at the screening examination (including laboratory tests and ECG).
* Screening ECG which demonstrates at least one of the following: heart rate > 100 bpm, QRS > 120 msec, QTc > 450 msec, PR > 220 msec or any rhythm other than sinus rhythm, sinus bradycardia, or sinus arrhythmia.
* Change in weight > 5 kilograms within 3 months of screening.
* History of alcohol consumption exceeding 14 drinks/week (1 drink equaling 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor) within the 6 months before study entry.
* Sitting systolic blood pressure ≤90 millimeters of mercury (mmHg) or ≥140 mmHg, diastolic blood pressure </= 50 mmHg or >/= 90 mmHg and judged to be clinically significant by the investigator.
* Positive result on drug screen, hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or human immunodeficiency (HIV) tests.
* Use of prescription or non-prescription drugs, vitamins, or dietary supplements within 14 days prior to the first dose of study medication. Subjects on oral contraceptives and subjects who have used acetaminophen at doses of < 2 grams/day are eligible for study entry. Any exception to this must be felt not to impact the integrity of the data and must be jointly agreed upon by the investigator and medical monitor.
* Treatment with any investigational drug, use of any known CYP450 enzyme- inducing/inhibiting agents (e.g., barbiturates, phenothiazines, cimetidine, St. John's Wort) or herbal supplements within 30 days prior to the first dose of study medication.
* Treatment with any psychotropic medication within 90 days of screening.
* History of drug abuse or dependence within 180 days of screening.
* Febrile illness within 5 days prior to the first dose of study medication.
* Inadequate venous access.
* Known allergy to sertraline or telenzepine.
* History of an active eating disorder such as anorexia nervosa, bulimia or binge eating disorder.
* Elevated ALT (> 2X ULN) or total bilirubin (> 1.6 mg/dL)
* Have diabetes mellitus (fasting plasma glucose > 126 mg/dL)
* Have been on weight loss medications in the past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Berg, MD, Principal Investigator — Cetero Research, San Antonio

RESULTS

PARTICIPANT FLOW:
Groups:
- Telenzepine - Group A: received Sertraline 0 mg/day for 7 days.After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
- Telenzepine Plus Sertraline - Group B: received Sertraline 50 mg/day for 7 days. After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
- Telenzepine Plus Sertraline - Group C: received Sertraline 100 mg/day for 7 days. After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
- Telenzepine Plus Sertraline - Group D: received Sertraline 150 mg/day for 7 days. After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
Period: Overall Study
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Telenzepine Plus Sertraline - Group C | Telenzepine Plus Sertraline - Group D
Started | 10 | 10 | 10 | 10
Completed | 9 | 10 | 8 | 9
Not Completed | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Telenzepine Plus Sertraline - Group C | Telenzepine Plus Sertraline - Group D | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Full Range); unit: years] | 30.7 [22 to 42] | 35.2 [21 to 45] | 33.5 [22 to 44] | 34.3 [22 to 45] | 33.4 [21 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 7 | 24
  Male | 5 | 5 | 3 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 7 | 6 | 26
  Not Hispanic or Latino | 3 | 4 | 3 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 2 | 9
  White | 8 | 6 | 7 | 8 | 29
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in the VAS Score From Baseline.
Description: The baseline VAS self-assessment was completed for each subject on day 7 of each dose combination. Appetite VAS was completed in the subject's room approximately 30 min before and 1 h after each meal serving. Appetite was not assessed prior to snacks. VAS assessment was based on response to the question: "How hungry are you now?" The anchor points of the 100mm scale were "I am not hungry at all" and "Never more hungry" corresponding to 0 mm and 100 mm respectively. The subjects' VAS scores were measured by the clinic staff and entered into the CRF. The description listed below (VAS after meal minus and VAS before meal) refers only to the mean VAS score of each group.
Time Frame: The baseline was defined on day 7 of sertraline treatment with no telenzepine before and meal. Appetite VAS was measured 30 min before and 1hour after to meal
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Telenzepine Plus Sertraline - Group B: received Sertraline 50 mg/day for 7 days.After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
- Sertraline Plus Telenzepine - Group C: received Sertraline 100 mg/day for 7 days.After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
- Sertraline Plus Telenzepine - Group D: received Sertraline 150 mg/day for 7 days.After 7 days, received telenzepine for 21 days total at 1, 2, and 3 mg/day for 7 days each.
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Sertraline Plus Telenzepine - Group C | Sertraline Plus Telenzepine - Group D
Number analyzed (Participants) | 10 | 10 | 10 | 10
mm
  1 mg of Telenzepine (30 min before breakfast) | 2.90 (28.77) | 2.70 (33.05) | -10.8 (25.72) | 6.70 (22.98)
  2 mg of Telenzepine (30 min before breakfast) | 5.50 (34.58) | -4.40 (24.80) | 18.50 (29.38) | -4.5 (32.74)
  3 mg of Telenzepine (30 min before breakfast) | 12.22 (34.66) | -7.60 (25.16) | 14.33 (31.86) | -4.60 (30.89)
  1 mg of Telenzepine (1 hour after breakfast) | 5.50 (16.64) | -2.40 (4.84) | -9.60 (40.56) | 1.20 (16.62)
  2 mg of Telenzepine (1 hour after breakfast) | 2.30 (8.18) | -5.20 (8.35) | 0.1 (20.90) | 6.70 (23.68)
  3 mg of Telenzepine (1 hour after breakfast) | 4.11 (13.01) | -7.60 (8.90) | -2.89 (31.85) | 3.50 (23.63)
  1 mg of Telenzepine (30 min before lunch) | 1.60 (18.76) | -14.50 (17.97) | -2.10 (26.21) | 4.60 (31.37)
  2 mg of Telenzepine (30 min before lunch) | -8.60 (23.32) | -16.30 (18.85) | 9.60 (24.47) | 2.40 (27.59)
  3 mg of Telenzepine (30 min before lunch) | -16.78 (25.37) | -23.40 (25.91) | 0.44 (21.90) | -2.70 (19.81)
  1 mg of Telenzepine (1 hour after lunch) | -2 (15.22) | -3.90 (15) | 4.60 (17.16) | 11 (23.32)
  2 mg of Telenzepine (1 hour after lunch) | -1.1 (12.34) | -6.10 (9.21) | 5.70 (7.90) | 2 (6.77)
  3 mg of Telenzepine (1 hour after lunch) | 0.44 (8.95) | -4.60 (8.91) | 12.11 (27.78) | 5.60 (22.37)
  1 mg of Telenzepine (30 min before supper) | -4.10 (30.35) | -1.20 (21.87) | 9.90 (26.41) | 12.50 (17.18)
  2 mg of Telenzepine (30 min before supper) | -14.10 (19.55) | -10.60 (17.05) | 4.50 (26.73) | 12.60 (21.61)
  3 mg of Telenzepine (30 min before supper) | -20.67 (37.51) | -17 (23.05) | -13.33 (30.64) | -1 (12.46)
  1 mg of Telenzepine (1 hour after supper) | 1.70 (7.57) | -3.10 (16.39) | -17 (8.38) | 13.70 (19.15)
  2 mg of Telenzepine (1 hour after supper) | 1.10 (7.78) | -3.30 (15.58) | -7 (17.33) | -3.30 (26.19)
  3 mg of Telenzepine (1 hour after supper) | -0.78 (3.93) | -4.30 (14.44) | -6.33 (16.65) | -8.10 (26.44)

2. Primary Outcome: Changes in the Meal Calories Consumed
Description: The changes in the meal calories consumed was measured upon telenzepine treatment at the dose of 1 mg, 2 mg and 3 mg (i.e. end of every 7 days). The baseline was defined as on day 7 of sertraline treatment with no telenzepine for the specified meal. Food consumption was measured as calories consumed for breakfast, lunch, and dinner for all treatment groups on day 7 of each dose combination.
Time Frame: The baseline was defined as on day 7 of sertraline treatment with no telenzepine. Food consumption was measured as calories consumed for breakfast, lunch, and dinner for all treatment groups on day 7 of each dose combination.
Measure: Mean (Standard Deviation); unit: calorie
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Sertraline Plus Telenzepine - Group C | Sertraline Plus Telenzepine - Group D
Number analyzed (Participants) | 10 | 10 | 10 | 10
calorie
  1 mg telenzepine (breakfast) | -63.70 (76.50) | -42.32 (144.91) | -88.93 (99.56) | -53.91 (125.23)
  2 mg telenzepine (breakfast) | 36.32 (82.34) | 23.70 (133.16) | -2.32 (78.06) | -67.36 (147.20)
  3 mg telenzepine (breakfast) | 58.59 (119.04) | 80.21 (170.09) | 68.21 (107.49) | -28.81 (144.40)
  1 mg telenzepine (lunch) | 13.98 (75.12) | 14.32 (66) | 59.69 (107.11) | 60.92 (91.62)
  2 mg telenzepine (lunch) | 33.91 (91.76) | 58.39 (129.87) | 144.50 (131.55) | 12.09 (111.57)
  3 mg telenzepine (lunch) | -22.36 (171.6) | -119.01 (173.82) | 2.92 (110.29) | -4.94 (153.37)
  1 mg telenzepine (supper) | -19.92 (110.88) | 47.66 (62.55) | 87.01 (171.07) | -79.49 (126.90)
  2 mg telenzepine (supper) | -26.16 (129.51) | -20.85 (139.59) | -13.10 (182.34) | -12.21 (152.92)
  3 mg telenzepine (supper) | 9.26 (140.61) | 61.88 (107.28) | -22.98 (183.93) | 42.85 (107.91)

3. Primary Outcome: Safety of Sertraline and Telenzepine Combination
Description: safety of the drug combination was measured in terms of number of adverse events during the study period.
Time Frame: 7 days
Measure: Number; unit: number of adverse events
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Sertraline Plus Telenzepine - Group C | Sertraline Plus Telenzepine - Group D
Number analyzed (Participants) | 10 | 10 | 10 | 10
number of adverse events
  Total | 10 | 17 | 25 | 47
  Mild | 9 | 15 | 20 | 43
  Moderate | 1 | 2 | 4 | 4
  Severe | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Telenzepine - Group A | Telenzepine Plus Sertraline - Group B | Telenzepine Plus Sertraline - Group C | Telenzepine Plus Sertraline - Group D
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 9/10 | 8/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telenzepine - Group A (N=10) | Telenzepine Plus Sertraline - Group B (N=10) | Telenzepine Plus Sertraline - Group C (N=10) | Telenzepine Plus Sertraline - Group D (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Head ache (Nervous system disorders) | 0 (0) | 5 (6) | 3 (3) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Increased urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Elevated fasting glucose (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes